CLINICAL TRIAL: NCT00260429
Title: Double-blind, Randomized Placebo Controlled Study of the Relative Safety and Efficacy of Collagenase Therapy in the Treatment of Residual-type Dupuytren's Disease.
Brief Title: Collagenase in the Treatment of Dupuytrens Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Biospecifics Technologies Corp. (Industry); Endo Pharmaceuticals (Industry)
Responsible Party: James Tursi, MD; VP of Clinical Development, Auxilium Pharmaceuticals, Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DUPY 303
Record Dates: First submitted 2005-11-29; First posted 2005-12-01 (Estimated); Results first posted 2010-12-09 (Estimated); Last update posted 2010-12-09 (Estimated); Status verified 2010-11

CONDITIONS: Dupuytren's Disease
Keywords: Dupuytren's contracture; fixed flexion contracture
MeSH Terms: conditions — Dupuytren Contracture | interventions — Microbial Collagenase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AA4500 0.58 mg (Experimental)
  Interventions: Biological: collagenase clostridium histolyticum
- placebo (Placebo Comparator)
  Interventions: Biological: collagenase clostridium histolyticum

INTERVENTIONS:
Biological: collagenase clostridium histolyticum — Subjects could have received up to three injections of AA4500/placebo into the cord of the affected hand. Each injection was separated by at least 30 days. Individual cords may have received up to a maximum of three injections.
  Other Names: XIAFLEX®; AA4500

SUMMARY:
The purpose of the study is to determine if collagenase will reduce the degree of contracture in the primary joint in subjects with Dupuytren's disease.

This study was designed to be part of the larger clinical program, for adult patients with Dupuytren's contracture with a palpable cord, where the data from 2 pivotal Placebo-Controlled studies (AUX-CC-857 and AUX-CC-859) and 7 non-pivotal studies were evaluated.

DETAILED DESCRIPTION:
In a random, placebo controlled, double blind study, collagenase injection therapy will be investigated for it's ability to disrupt the Dupuytren's cord.

Resultant cord disruption may obviate the need for patients to have surgery to correct the finger flexion contractures of Dupuytren's disease.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were at least 18 years of age, of either sex or any race.
* Subjects had residual Dupuytren's disease with a fixed-flexion deformity of the finger(s) of at least 20 degrees or greater, caused by a palpable cord.
* Subjects had a positive "table-top test" defined as the inability to simultaneously place their affected finger(s) and palm flat against a table top.
* Subjects must have been willing to participate in and complete the study, and comply with its procedures by signing an IRB approved written consent form.
* Subjects must have been able to understand and adhere to the visit schedule. They must have been able to follow study procedures and instructions, and have agreed to report concomitant medications and adverse events accurately and consistently.
* Women of childbearing potential must have agreed to use an acceptable method of birth control or must have been surgically sterilized (hysterectomy or tubal ligation). Women of childbearing age had a urine pregnancy test on Day 0 (day of injection) prior to the injection.

Exclusion Criteria

* Women who were nursing or who were pregnant (as evidenced by a positive urine pregnancy test at the time of enrollment).
* Subjects who had participated in an investigational drug trial within 30 days of enrollment in this study.
* Subjects who had received surgery for Dupuytren's disease within 30 days of enrollment in this study.
* Subjects who had a known allergy to AA4500 or any of the inactive ingredients in the AA4500 injection.
* Subjects who had a known allergy to doxycycline.
* Subjects who had a medical condition that would have made them unsuitable for enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-06; Primary Completion 2005-08 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence C Hurst, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital and Mediacl Center, Stony Brook, New York, United States

REFERENCES:
- [Background] Badalamente MA, Hurst LC, Hentz VR. Collagen as a clinical target: nonoperative treatment of Dupuytren's disease. J Hand Surg Am. 2002 Sep;27(5):788-98. doi: 10.1053/jhsu.2002.35299. PMID 12239666
- See also: XIAFLEX Prescribing Information — http://www.accessdata.fda.gov/drugsatfda_docs/label/2010/125338lbl.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- AA4500: collagenase clostridium histolyticum 0.58mg injected into metacarpophalangeal (MP) and/or proximal interphalangeal (PIP) joints
Period: Overall Study
Arm/Group | AA4500 | Placebo
Started | 23 | 12
Completed | 21 | 12
Not Completed | 2 | 0
Not completed — failure to follow appointments | 1 | 0
Not completed — scheduled hand surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AA4500 | Placebo | Total
Number analyzed (Participants) | 23 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 5 | 21
  >=65 years | 7 | 7 | 14
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (7.6) | 63.8 (10.0) | 61.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 20 | 8 | 28
Region of Enrollment [Number; unit: participants]
  United States | 23 | 12 | 35

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure is Reduction of Flexion Contracture of the Primary Joint.
Description: The Primary Outcome Measure for patients treated with AA4500 is the percentage of 23 joints that were successfully treated where "successfully treated" was defined as reduction in contracture to 5° or less.
  The Primary Outcome Measure for placebo treated patients is the percentage of 12 joints that were successfully treated where "successfully treated" was defined as reduction in contracture to 5° or less.
Time Frame: 30 days after the last injection
Measure: Number; unit: % Joints
Arm/Group | AA4500 | Placebo
Number analyzed (Participants) | 23 | 12
% Joints | 91.3 | 0

2. Secondary Outcome: Percent Reduction From Baseline Contracture After the Last Injection
Time Frame: 30 days after last treatment to the primary joint
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Joints

3. Secondary Outcome: Percent Change From Baseline Range of Motion After the Last Injection
Time Frame: 30 days after last treatment to the primary joint
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: Joints

4. Secondary Outcome: Time to First Achieve and Maintain Clinical Success After the Last Injection
Time Frame: First evaluation visit on which clinical success is achieved and maintained through the Day 30 evaluation of the primary joint
Reporting Status: Not Posted
Measure: Number; unit: Joints

5. Secondary Outcome: Clinical Success After the First Injection
Time Frame: 30 days after first treatment to the primary joint
Reporting Status: Not Posted
Measure: Number; unit: Joints

6. Secondary Outcome: Percent Reduction From Baseline Contracture After the First Injection
Time Frame: 30 days after first treatment to the primary joint
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Joints

7. Secondary Outcome: Change From Baseline Range of Motion After the First Injection
Time Frame: 30 days after first treatment to the primary joint
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Joints

ADVERSE EVENTS:
Description: This study was designed to be part of the larger clinical program. For information regarding XIAFLEX-associated Serious and Non-serious Adverse events please refer to the XIAFLEX Medication Guide & XIAFLEX Prescribing Information (see links above).
Arm/Group | AA4500 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/23 | 1/15
Other Adverse Events (participants affected / at risk) | 23/23 | 12/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | AA4500 (N=23) | Placebo (N=15)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0/12 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1/12 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AA4500 (N=23) | Placebo (N=15)
Edema peripheral (General disorders) | 23 | 1
Injection site pain (General disorders) | 23 | 7
Ecchymosis (Skin and subcutaneous tissue disorders) | 12 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 10 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 10 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 0
Tenderness (General disorders) | 3 | 0
Body temperature increased (Investigations) | 2 | 0
Headache (Nervous system disorders) | 2 | 0
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3
Hypertension (Vascular disorders) | 1 | 2
nasopharyngitis (Infections and infestations) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes